CLINICAL TRIAL: NCT02697877
Title: Assessment and Prognostic Significance of Global Myocardial Perfusion Reserve Using Coronary Sinus Flow Measurements During Regadenoson Stress Cardiac Magnetic Resonance
Brief Title: Assessment of Global Myocardial Perfusion Reserve Using Coronary Sinus Flow Measurements
Status: Completed | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Afshin Farzaneh-Far, Assistant Professor of Clinical Medicine, University of Illinois at Chicago
Other Study IDs: 2015-1275
Record Dates: First submitted 2016-02-24; First posted 2016-03-03 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — regadenoson

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with known or suspected coronary artery disease.: Patients with known or suspected coronary artery disease undergoing clinically ordered stress cardiac magnetic resonance imaging.
  Interventions: Drug: Regadenoson

INTERVENTIONS:
Drug: Regadenoson

SUMMARY:
The aim of this study is to assess whether myocardial perfusion reserve, measured during routine clinically ordered regadenoson stress cardiac magnetic resonance (CMR) has prognostic value in predicting adverse cardiovascular events. Myocardial perfusion reserve will be measured with CMR by assessing blood flow through the coronary-sinus - the primary vein in the heart.

DETAILED DESCRIPTION:
Myocardial perfusion reserve is the ratio of global myocardial blood flow at stress vs. rest. Traditionally, it has been measured non-invasively using quantitative positron emission tomography (PET) or cardiac magnetic resonance (CMR). Several recent studies have suggested that measurement of myocardial perfusion reserve provides significant additive prognostic information during stress perfusion imaging in patients with known or suspected coronary artery disease. Myocardial perfusion reserve depends not only on trans-stenotic pressure gradient of the epicardial arteries and thus stenosis severity but even more on the ability of the coronary microvasculature (especially the pre-arterioles) to dilate. Therefore, coronary microvascular dysfunction, which impairs pre-arteriolar function, reduces myocardial perfusion reserve independently of the presence of epicardial coronary stenosis. Hence, the ability to measure myocardial perfusion reserve allows a more comprehensive assessment of the entire coronary circulation, beyond the current paradigm of the epicardial arteries.

However, both PET and current CMR techniques are cumbersome, and in the case of PET require radiation as well as on-site Rubidium-82 generators. Therefore, they are challenging for routine clinical practice and have been limited to specialized research centers. An alternative, simple CMR method for measurement of myocardial perfusion reserve by quantifying change in coronary sinus flow has been described. The coronary sinus drains approximately 96% of total myocardial blood flow and provides a potentially convenient location for measurement of global myocardial blood flow. This method has been validated against both invasive and PET techniques. The investigators hypothesized that measurement of coronary sinus flow at stress and rest may provide a simple and rapid assessment of myocardial perfusion reserve during regadenoson stress perfusion CMR.

This study will use phase contrast images obtained from patients during their clinically indicated CMR stress study to calculate myocardial perfusion reserve as the ratio of maximum myocardial blood flow to baseline blood flow - at the coronary sinus. Coronary sinus flow will be calculated by post-processing of images after the patient has left the scanner. In brief, the contour of the coronary sinus will be traced on the flow images throughout the cardiac cycle. Coronary sinus flow is calculated by integrating the momentary flow rate values from each cardiac phase over the entire cardiac cycle and multiplying by the mean heart rate during the acquisition. Patients will be followed for the occurrence of major adverse cardiac events (death, myocardial infarction, late revascularization, hospitalization for heart failure or unstable angina).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Male or Female
* Referred for clinical cardiac magnetic resonance stress testing (with Regadenoson) at the University of Illinois Hospital & Health Sciences System by their healthcare provider as part of their routine clinical care for known or suspected coronary artery disease.

Exclusion Criteria:

* Presence of metallic implants contraindicated with cardiac magnetic resonance (e.g. implantable cardiac defibrillator, pacemaker)
* Glomerular Filtration Rate (GFR) <30ml/min
* High degree atrio-ventricular block
* Hypersensitivity to Regadenoson
* Severe active wheezing from asthma
* Severe claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18yrs who are undergoing clinically indicated stress cardiac magnetic resonance (CMR) imaging for known or suspected coronary artery disease.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2016-02; Primary Completion 2018-02 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events | For upto 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- 1740 W Taylor Street, 2nd Floor, Cardiac Imaging, Chicago, Illinois, United States